CLINICAL TRIAL: NCT03663634
Title: Cytochalasin B Supplementation to ICSI Handling Medium
Brief Title: Supplementing Intracytoplasmic Sperm Injection Handling Medium With Cytochalasin B
Acronym: ICSI-CB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Sina Hospital (Other Government)
Collaborators: Banoon IVF Center (Other)
Responsible Party: Principal Investigator, Muhammad Fawzy, IVF Lab Director, Ibn Sina Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IbnSinaIVF-ICSI-CB
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Handling Medium Supplemented with Cytochalasin B (Experimental)
  Interventions: Other: Cytochalasin B use in ICSI handling medium
- Handling Medium as it is. (No Intervention)

INTERVENTIONS:
Other: Cytochalasin B use in ICSI handling medium — A medium with in-house supplementation of Cytochalasin B to decrease oocyte degeneration after ICSI and improve survival rate
  Arms: Handling Medium Supplemented with Cytochalasin B

SUMMARY:
Vienna Consensus has identified 10% damage rate after ICSI as a competency value. Despite the highest quality embryologists doing ICSI, degeneration sometimes occurs due to oocyte factors such as the fragile membrane, etc. Cytochalasin B serves to facilitate spindle or pronuclear transfer procedures helping to reduce the damage rate with no harm reported. Using Cytochalasin B during ICSI could serve to rescue some oocytes from the degeneration allowing for more chances of viable zygotes,

ELIGIBILITY:
Inclusion Criteria:

* All ICSI candidates patients

Exclusion Criteria:

* No exclusion

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 987 (Actual)
Dates: Start 2018-09-16 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
oocyte survival rate | 6 days of culture
  number of survived oocyte after intracytoplasmic sperm injection

SECONDARY OUTCOMES:
fertilization rate | 6 days of culture
  number of fertilized oocytes per metaphase II injected
blastocyst formation rate | 6 days of culture
  number of formed blastocyst per fertilized oocyte
embryo utilization rate | 6 days of culture
  number of embryo transferred added to number of those cryopreserved per fertilized oocyte
clinical pregnancy rate | three months
  number of women with a heartbeat at week 4 or more after embryo transfer
ongoing pregnancy rate | four months
  number of women with continued pregnancy after twelve weeks of gestation

CONTACTS AND LOCATIONS:
Locations (1):
- IbnSina IVF Center, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No